CLINICAL TRIAL: NCT04633759
Title: Feasibility of Low-load Resistance Training Using Blood Flow Restriction for People With Multiple Sclerosis and Marked Mobility Restriction
Brief Title: Low Load Resistance Training Using Blood Flow Restriction for People With Multiple Sclerosis
Acronym: BFR-MS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Consortium of Multiple Sclerosis Centers (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-0695; 205593 (Other Grant/Funding Number: Consortium of Multiple Sclerosis Centers)
Record Dates: First submitted 2020-11-12; First posted 2020-11-18 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Blood Flow Restriction; Resistance Training
MeSH Terms: conditions — Multiple Sclerosis | interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Blood Flow Restriction Exercise (Experimental): Participant will participate in a supervised low load blood flow restriction exercise program twice a week for 8 weeks.
  Interventions: Other: Blood Flow Restriction Exercise

INTERVENTIONS:
Other: Blood Flow Restriction Exercise — Following a 5-minute low intensity warm-up, the BFR cuff will be placed at the most proximal portion of the leg and dosed following standard BFR guidelines: 1 set of 30 reps, then 3 sets of 15 reps at 20-30% 1RM with up to 80% limb occlusion. Exercises will target bilateral 1) knee and hip extension, 2) hip abduction, and 3) ankle plantarflexion, as these muscles are important for functional mobility in people with MS.

SUMMARY:
The Primary Aim of this research study is to determine the feasibility of 8 weeks of physical therapy strengthening exercises using blood flow restriction (BFR) in people with multiple sclerosis (MS) who have moderate-to-severe walking problems. BFR training involves placing a cuff on the leg being exercised in order to restrict blood flow. The cuff is attached to a specialized device that automatically detects the appropriate amount of pressure to place on the limb. Testing will occur before and after the 8-week treatment period.

DETAILED DESCRIPTION:
The Primary Aim of this research study is to determine the feasibility of 8 weeks of physical therapy strengthening exercises using blood flow restriction (BFR) in people with multiple sclerosis (MS) who have moderate-to-severe walking problems. BFR training involves placing a cuff on the leg being exercised in order to restrict blood flow. The cuff is attached to a specialized device that automatically detects the appropriate amount of pressure to place on the limb. Testing will occur before and after the 8-week treatment period.

Specific Aim 1: Determine the feasibility of BFR by assessing recruitment rate, retention, adherence, satisfaction, and safety.

Hypothesis: Feasibility will be demonstrated by: 1) enrolling 20 participants in 8 months, 2) retaining at least 16 (80%) participants, 3) 80% adherence to intervention, 4) 90% satisfaction with intervention, and 5) no serious adverse events related to the intervention.

Specific Aim 2: Determine changes in knee and hip extension, hip abduction, and ankle plantarflexion muscle strength after the 8-week intervention.

Hypothesis: Following intervention there will be clinically important within-group strength changes that correspond to established minimal detectable change values and which can be characterized as having at least a moderate effect size as defined by Cohen's d.

Exploratory Aim: Explore changes in functional mobility (30-Second Sit-to-Stand, Berg Balance Scale, Timed 25-Foot Walk. 10-day average activity level) and self-report measures (12-Item MS Walking Scale, Modified Fatigue Impact Scale, MS Impact Scale-29, and Patient-Specific Functional Scale) after the 8-week intervention.

ELIGIBILITY:
Inclusion Criteria:

* Adults ages 18-70
* Neurologist-confirmed diagnosis of multiple sclerosis
* Expanded Disability Status Scale (EDSS) 6.0 to 7.0

  * EDSS 6.0: unilateral assistance (cane or crutch) required to walk at least 100 meters with or without resting
  * EDSS 6.5: Bilateral assistance (cane or crutch) required to walk at least 20 meters with or without resting
  * EDSS 7.0: unable to walk 5 meters even with aid, essentially restricted to wheelchair; wheels self and transfers alone; up and about in wheelchair some 12 hours a day

Exclusion Criteria:

* EDSS 7.5 or greater: Restricted to wheelchair for all mobility, unable to walk more than a few steps, even with walking aid
* EDSS 5.5 or less: Able to walk more than 100 meters without walking aid or rest
* Unable to provide consent or follow simple directions
* Prior history of Deep Venous Thrombosis/ Pulmonary Embolism
* History of peripheral vascular disease, thrombophilia or other clotting disorders
* Patient report of easy bruising
* Any comorbid conditions or pain that substantially affects physical function or would interfere with the participant's ability to safely complete rehabilitation (e.g. neurologic, vascular, cardiac problems, orthopedic, or ongoing medical treatments) as determined by a neurologist of physical therapist
* Severe lower extremity spasticity as defined as Modified Ashworth scale > 2
* Currently undergoing supervised resistance training with a physical therapist or other exercise professional
* Use of Blood Flow Restriction currently or in the previous 3 months prior to enrollment
* MS-related exacerbation or changes to their disease-modifying drug therapy in the month prior to enrollment
* Inability to tolerate pressure cuff during baseline assessment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-02-19 (Actual); Primary Completion 2022-10-05 (Actual); Study Completion 2022-10-05 (Actual)

PRIMARY OUTCOMES:
Change in knee extension muscle strength | Measured at Baseline (Week 0) and Post Test (Week 9)
  Knee extension muscle strength measured by hand-held dynamometry
Change in hip abduction muscle strength | Measured at Baseline (Week 0) and Post Test (Week 9)
  Hip abduction muscle strength measured by hand-held dynamometry
Change in ankle plantarflexion muscle strength | Measured at Baseline (Week 0) and Post Test (Week 9)
  Ankle plantarflexion muscle strength measured by hand-held dynamometry

SECONDARY OUTCOMES:
Change in 30-second sit-to-stand completions | Measured at Baseline (Week 0) and Post Test (Week 9)
  Functional mobility test measuring the number of sit to stand cycles a participant can complete in 30 seconds
Change in Berg Balance Scale | Measured at Baseline (Week 0) and Post Test (Week 9)
  Functional mobility test measuring the participant's ability to balance in different postures. Scores range from 0 to 56 points, with 0-20 points indicating wheelchair bound, 21-40 indicating walking with assistance, and 41-56 indicating walking independently.
Change in timed 25-foot walk | Measured at Baseline (Week 0) and Post Test (Week 9)
  Functional mobility test measuring the time it takes a participant to walk 25 feet
Change in activity level | Measured at Baseline (Week 0) and Post Test (Week 9)
  10-day average of activity level as measured by a wearable activity monitor
Change in 12-Item MS Walking Scale | Measured at Baseline (Week 0) and Post Test (Week 9)
  Self-report questionnaire measuring walking ability with scores ranging from 12 points (no difficulty walking, to 60 points (extremely limited or no walking)
Change in Modified Fatigue Impact Scale | Measured at Baseline (Week 0) and Post Test (Week 9)
  Self-report questionnaire measuring fatigue caused by MS with scores ranging from 0 (no impact of fatigue in the past 4 weeks) to 84 (maximum impact of fatigue in the past 4 weeks)
Change in MS Impact Scale-29 | Measured at Baseline (Week 0) and Post Test (Week 9)
  Self-report questionnaire measuring the impact of MS on daily activity with scores ranging from 29 (MS has no impact on my daily life) to 145 (MS extremely impacts my daily life)
Change in MS Patient-Specific Function Scale | Measured at Baseline (Week 0) and Post Test (Week 9)
  Self-report questionnaire measuring the ability of the participant to do three self-identified activities. Scores of each of the 3 activities range from 0 (unable to perform) to 10 (able to perform without difficulty)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado, Aurora, Colorado, United States

REFERENCES:
- [Derived] Manago MM, Cohen ET, Cameron MH, Christiansen CL, Bade M. Reliability, Validity, and Responsiveness of the Patient-Specific Functional Scale for Measuring Mobility-Related Goals in People With Multiple Sclerosis. J Neurol Phys Ther. 2023 Jul 1;47(3):139-145. doi: 10.1097/NPT.0000000000000439. Epub 2023 Mar 7. PMID 36897202